CLINICAL TRIAL: NCT05442229
Title: A Study to Establish the Norm of Chinese Speech and Language Development in Children Aged 2 ~ 6
Brief Title: A Cross-sectional Study to Evaluate Speech and Language Development in Chinese Children Aged 2-6 Years
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: WHTJYYLB
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-03

CONDITIONS: Mental Retardation; Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder
Keywords: language development; development assessment; speech and language assessment scale
MeSH Terms: conditions — Intellectual Disability; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Speech

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normally developing child: Normal development is defined as children without intellectual development disorders, developmental speech or language disorders, ASD (autism spectrum disorder), and ADHD (attention deficit hyperactivity disorder).
  Interventions: Other: establish a new Chinese children's speech and language norm
- Abnormally developed child: Abnormal development is defined as that hospital visits of children were professionally assessed for MR (mental retardation), ASD (autism spectrum disorder), and ADHD (attention deficit hyperactivity disorder). Diagnostic criteria were all referred to Diagnostic and Statistical Manual of Mental Disorders，DSM-5.
  Interventions: Other: establish a new Chinese children's speech and language norm

INTERVENTIONS:
Other: establish a new Chinese children's speech and language norm — 1063 normally developing children and 96 abnormally developing children will be retrospectively enrolled from the medical records of stratified, randomly selected centers. A total of 4137 children with normal development and 448 children with abnormal development aged from 2 to 6 years old will be selected from 11 hospitals in China by multi-center, stratified, unequal proportion random sampling and face-to-face survey. Children's speech and language development was assessed by the Speech and Language Development Scale for children aged 2 to 6, compiled by the Linguistics and Language Research Centre of the Education University of Hong Kong.

SUMMARY:
The purpose of this study is to establish a new Chinese children's speech and language norm by obtaining the latest data of speech and language development of children aged 2 ~ 6 from different regions in China. At the same time, the overall development level and group differences of speech and language in Chinese children aged 2 to 6 years, and the influencing factors of speech and language development in Chinese children aged 2 to 6 years were also discussed.

DETAILED DESCRIPTION:
1. To establish the norm of speech and language development in Chinese children aged 2 to 6 1063 normally developing children and 96 abnormally developing children will be retrospectively enrolled from the medical records of stratified, randomly selected centers. A total of 4137 children with normal development and 448 children with abnormal development aged from 2 to 6 years old will be selected from 11 hospitals in China by multi-center, stratified, unequal proportion random sampling and face-to-face survey. Children's speech and language development was assessed by the Speech and Language Development Scale for children aged 2 to 6, compiled by the Linguistics and Language Research Centre of the Education University of Hong Kong.
2. To investigate and analyze the present situation of speech and language development of children aged 2-6 in China The present situation of children's speech and language development was analyzed, and the differences of gender, age, birth and other influencing factors were statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

For normally developing children

1. All children must meet all of the following criteria simultaneously:
2. Informed consent of legal guardian or group representative;
3. Age from 2 to 6 years old, male and female;
4. Native speaker of Mandarin;
5. Children in kindergartens and hospitals are professionally assessed as normal development, which is defined as children without intellectual development disorder, developmental speech or language disorder, autism spectrum disorder, and attention deficit hyperactivity disorder.

   For abnormally developed children
6. Informed consent of legal guardian or group representative;
7. Age from 2 to 6 years old, male and female;
8. Native speaker of Mandarin;
9. Children with intellectual development disorder, autism spectrum disorder and attention deficit hyperactivity disorder are assessed professionally in the hospital; Diagnostic criteria were referred to Diagnostic and Statistical Manual of Mental Disorders (DSM-5)

Exclusion Criteria:

For normally developing children

1. Poor coordination;
2. Other unsuitable children considered by researchers, such as children whose developmental level is basically normal but whose environmental and socio-economic factors (premature birth, low birth weight, malnutrition, abuse, etc.) have been verified to affect language development.

   For abnormally developed children
3. Study the poor fit degree;
4. Have visual and hearing impairment;
5. Other unsuitable children considered by researchers, such as children with other organic dysfunction, such as cerebral palsy, congenital genetic diseases, epilepsy, etc.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2 to 6 years of normal and abnormal development of children in 11 hospitals in China (covering central, east, South, west, North and east China) North area) and the corresponding area of the kindergarten
Sampling Method: Probability Sample
Enrollment: 5744 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Chinese children's speech and language norm | 2021.11.1-2023.5.1
  The speech and Language Development Scale for children aged 2 to 6 was developed by the Linguistics and Language Research Center of the Education University of Hong Kong. It was divided into three parts: phonological assessment (word pronunciation), vocabulary assessment (comprehension and expression) and grammar assessment (comprehension). Color hand-painted pictures were used for the evaluation of the three types of items, and words were named by pictures, and words were selected by listening and listening, so as to ensure the practicality and conciseness of the scale, as well as the simplicity of operation and implementation. Finally, the total score of each subject was calculated and relevant developmental status conclusions were drawn.